CLINICAL TRIAL: NCT06692725
Title: De-escalation of Neoadjuvant Chemotherapy Regimens (Taxane Plus Carboplatin Versus Taxane Plus Carboplatin Sequential Anthracycline) With Immunotherapy Among TNBC
Brief Title: De-escalation of Neoadjuvant Chemotherapy Regimens With Immunotherapy Among TNBC
Acronym: NacTNBC
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Other Study IDs: PKUPH2024Z160
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Triple Negative Breast Cancer
Keywords: neoadjuvant chemotherapy; De-escalation
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumor paraffin sample for each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Taxanes combined with carboplatin sequential anthracycline: Paclitaxel, liposome paclitaxel, docetaxel, or albumin paclitaxel combined with carboplatin for 4 cycles, followed by anthracycline combined with cyclophosphamide for 4 cycles, and PD-1 inhibitor was used at the same time
- Taxanes combined with carboplatin: paclitaxel, liposome paclitaxel, docetaxel, or albumin paclitaxel combined with carboplatin for 6 cycles, and PD-1 inhibitor was used at the same time

SUMMARY:
The traditional neoadjuvant therapy for triple negative breast cancer is based on anthracycline, paclitaxel and carboplatin. Nowadays, immunotherapy combined with chemotherapy has become a new standard treatment, which not only benefits from pathological complete response (pCR), but also benefits from long-term survival. The standard chemotherapy combined with immunotherapy scheme recommended by the guidelines is TCb-AC combined with pabolizumab, but the complex chemotherapy scheme has the defects of long cycle and large adverse reactions, and the scheme of chemotherapy reduction has been explored.

This project plans to adopt an ambispective cohort study, based on the large sample breast disease cohort database established by the breast center of Peking University People's Hospital, and retrospectively include the triple negative breast cancer patients with clinical stage T2 and above and/or lymph node positive who received neoadjuvant therapy (TCb-AC combined with immunotherapy, or TCb combined with immunotherapy) admitted to the center from January 1, 2019 to November 31, 2024. Patients of the same type from December 1, 2024 to December 31, 2028 were prospectively included. The efficacy and safety of different treatment regimens were compared.

DETAILED DESCRIPTION:
Investigators retrospectively recruited the triple negative breast cancer patients with clinical stage T2 and above and/or lymph node positive who received neoadjuvant therapy (TCb-AC combined with immunotherapy, TCb combined with immunotherapy, or TCb chemotherapy only) admitted to the center from January 1, 2019 to November 31, 2024. Patients of the same type from December 1, 2024 to December 31, 2028 were prospectively included. The efficacy and safety of different treatment regimens were compared.

Inclusion Criteria:

1. Patients with triple negative breast cancer diagnosed by biopsy in Peking University People's Hospital;
2. The clinical stage was stage II or stage III (i.e. T2 and above, and/or lymph node positive, without distant organ metastasis);
3. Received treatment in our hospital and had hospitalization records;
4. Has signed and agreed to participate in the PKUPH breast disease cohort study.

Exclusion Criteria:

1. Lack of clinical and pathological data (such as imaging data and pathological data);
2. Patients with metastatic breast cancer or bilateral breast cancer;
3. At the same time, they received anti-tumor therapy in other clinical trials, including endocrine therapy and targeted therapy;
4. Receiving other regimens besides the established neoadjuvant regimens

Primary end point: pathology complete response

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with triple negative breast cancer diagnosed by biopsy in Peking University People's Hospital;
* 2) The clinical stage was stage II or stage III (i.e. T2 and above, and/or lymph node positive, without distant organ metastasis);
* 3) Received treatment in our hospital and had hospitalization records;
* 4) Has signed and agreed to participate in the PKUPH breast disease cohort study.

Exclusion Criteria:

* 1) Lack of clinical and pathological data (such as imaging data and pathological data);
* 2) Patients with metastatic breast cancer or bilateral breast cancer;
* 3) At the same time, they received anti-tumor therapy in other clinical trials, including endocrine therapy and targeted therapy;
* 4) Receiving other regimens besides the established neoadjuvant regimens

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: triple negative breast cancer patients who received neoadjuvant chemotherapy based on taxanes combined with carboplatin
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
pathology complete response | 6 months
  Postoperative pathology confirmed that the primary breast lesions and axillary lymph nodes had no residual invasive tumor cells (ypT0/is and ypN0)

SECONDARY OUTCOMES:
Invasive disease free survival | 5 years
  the time from study enrollment to the first occurrence of the following events defined as failure: local recurrence of ipsilateral invasive breast cancer, contralateral invasive breast cancer, distant recurrence or death from any cause.
Disease free survival | 5 years
  the time from study enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause.
Breast cancer specific survival | 5 years
  time from study enrollment to death due to breast cancer.
Overall survival | 5 years
  the time from study enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: shu wang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China